CLINICAL TRIAL: NCT05813691
Title: Epidemiology of Occult Hepatitis C Virus Infection in Patients Born Before 1969 in the Hospital Setting: a Spontaneous Opportunistic Screening Initiative.
Acronym: ERADIcATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Ponziani Francesca Romana, Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5494
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C, Chronic; Hepatitis C; Hepatitis
Keywords: hepatitis C virus
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Meridan Bioscience Point of Care test against HCV antibodies — Point of care evaluation of antibodies against HCV obtaining a drop of capillary blood via puncture of the fingertip. If antibodies were detected, HCV RNA assay will be performed.

SUMMARY:
The goal of this monocentric prospective observational study is to evaluate the prevalence of unknown hepatitis C virus chronic infection in general population born before january 1st 1968 in Italy.

The main questions it aims to answer are:

what is the prevalence of hepatits C virus infection in general population born before January 1st, 1968? What rare the characteristics of these patients compared to the general population? What is the prevalence of patients tested HCV positive who are referred to the Hepatology Outpatient Clinic for further evaluation? What is the prevalence of patients with HCV infection detected during the study and treated with direct antiviral agents during follow up?

Participants will be tested with a point of care screening test (Meridian, Bioscience) able to detect anti-HCV antibodies to detect the presence of antibodies against HCV.

ELIGIBILITY:
Inclusion Criteria:

* Patients born before January 1st 1968 who lived in Italy referred to any departments of the Policlinico A. Gemelli

Exclusion Criteria:

* Patients born after january 1st 1968
* Known infection of hepatitis C virus
* Previous treatment against hepatitis C virus

Ages: 54 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients born before January 1st 1968 who lived in Italy referred to any departments of the Policlinico A. Gemelli
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of antibodies against hepatitis C virus in cohort population | 24 months
  Evaluation of prevalence of antibodies against HCV in patients referred to any department of Policlinico Gemelli born before January 1st 1968

SECONDARY OUTCOMES:
Characteristics of population | 24 months
Prevalence of patients with a confirmed chronic HCV infection who are referred to Hepatology Outpatient clinic | 24 months
Prevalence of patients with a confirmed chronic HCV infection who are treated with direct antiviral agents | 24 months